CLINICAL TRIAL: NCT06064097
Title: A Phase 2 Study Using Chemoimmunotherapy With Gemcitabine, Cisplatin and Nivolumab in Newly Diagnosed Nasopharyngeal Carcinoma (NPC)
Brief Title: A Study Using Nivolumab, in Combination With Chemotherapy Drugs to Treat Nasopharyngeal Carcinoma (NPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-07208; NCI-2023-07208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARAR2221 (Other: Children's Oncology Group); ARAR2221 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2023-09-29; First posted 2023-10-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Stage II Nasopharyngeal Carcinoma AJCC v8; Stage III Nasopharyngeal Carcinoma AJCC v8; Stage IV Nasopharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Biopsy; Specimen Handling; X-Rays; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; fluciclovine F-18; Gemcitabine; Magnetic Resonance Spectroscopy; Nivolumab; Radiotherapy; Radiation; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nivolumab, gemcitabine, cisplatin, radiation) (Experimental): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Chest Radiography; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Echocardiography Test; Other: Electronic Health Record Review; Other: Fluciclovine F18; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Other: Electronic Health Record Review — Ancillary studies
Other: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Receive radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: X-Ray Imaging — Undergo dental x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial tests effects of nivolumab in combination with chemotherapy drugs prior to radiation therapy patients with nasopharyngeal carcinoma (NPC). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Researchers want to find out what effects, good and/or bad, adding nivolumab to chemotherapy has on patients with newly diagnosed NPC. In addition, they want to find out if children with NPC may be treated with less radiation therapy and whether this decreases the side effects of therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate safety of combining chemotherapy (cisplatin and gemcitabine) with an anti-PD1 immune checkpoint inhibitor (nivolumab) in children, adolescents and young adults with nasopharyngeal carcinoma (NPC) by determining the rate of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher immune related adverse events (irAEs).

SECONDARY OBJECTIVES:

I. To estimate the 2-year event-free survival (EFS) of children, adolescents and young adults with NPC who are treated with induction chemoimmunotherapy (CIT), followed by consolidation chemoradioimmunotherapy (CRIT, cisplatin, nivolumab and response-adjusted, dose de-escalated radiation therapy), and nivolumab maintenance therapy.

II. To evaluate the objective response rate (ORR) including complete responders and partial responders (complete response [CR] + partial response [PR]) of neoadjuvant CIT.

III. To evaluate feasibility of combining chemotherapy (cisplatin and gemcitabine) with an anti-PD1 immune checkpoint inhibitor (nivolumab) in children, adolescents and young adults with nasopharyngeal carcinoma (NPC).

IV. To evaluate the cumulative incidence of local and distant relapse.

EXPLORATORY OBJECTIVES:

I. To estimate 5-year EFS and overall survival (OS) of children with NPC who are treated with induction CIT followed by consolidation CRIT, and nivolumab maintenance therapy.

II. To compare response assessed by fludeoxyglucose F18 (FDG) positron emission tomography (PET) versus magnetic resonance imaging (MRI).

III. To determine treatment outcomes for patients treated with radiation per protocol versus (vs) deviation.

IV. To evaluate outcomes comparing patients receiving intensity modulated radiation therapy (IMRT) to proton therapy.

V. To objectively measure both acute and long-term toxicity including immune related adverse events and radiation late effects.

VI. To evaluate swallowing dysfunction using patient reported outcome (PRO) measures for children and adults throughout the protocol for up to 5 years.

VII. To evaluate quality of life (QOL) using Patient-Reported Outcomes Measurement Information System (PROMIS) multidimensional questionnaire throughout the protocol for up to 5 years.

VIII. To correlate the lymphocyte to monocyte ratio on complete blood counts (CBCs) with treatment response and outcomes.

IX. To collect and bank specimens (including tumor, blood and stool) for future research studies.

OUTLINE:

INDUCTION THERAPY: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle, gemcitabine IV over 30 minutes on days 1 and 8 of each cycle, and cisplatin IV over 3-6 hours on day 1 of each cycle. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY: Patients receive nivolumab IV over 30 minutes on day 1 of each cycle and cisplatin IV over 3-6 hours on day 1 of cycles 1-2. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive concurrent radiation therapy on trial.

MAINTENANCE THERAPY: Patients receive nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening and as clinically indicated on trial. Patients undergo MRI, FDG PET, and computed tomography (CT) throughout the trial and chest x-ray during follow-up. Patients also undergo dental x-ray imaging on the trial. Patients may optionally undergo tissue biopsy, blood and stool sample collection during screening and on trial.

After completion of study treatment, patients are followed up every 3 months for 12 months, every 6 months until 24 months off therapy, and then yearly until 5 years off therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≤ 21 years of age at the time of study enrollment
* Newly diagnosed American Joint Committee on Cancer (AJCC) stage II-IV nasopharyngeal carcinoma (NPC)

  * Patients must have had histologic verification of the malignancy at original diagnosis
  * Although submission of tumor tissue for the molecular characterization initiative is not required for eligibility, it is strongly recommended
* Patients must have had histologic verification of the malignancy at original diagnosis
* Although submission of tumor tissue for the molecular characterization initiative is not required for eligibility, it is strongly recommended
* Patients must have a Lansky (for patients ≤ 16 years of age) or Karnofsky (for patients > 16 years of age) performance status score of ≥ 60%
* Peripheral absolute neutrophil count (ANC) ≥ 1000/uL (within 7 days prior to start of protocol therapy)
* Platelet count ≥ 100,000/uL (transfusion independent) (within 7 days prior to start of protocol therapy)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2 or (within 7 days prior to start of protocol therapy)
* A serum creatinine based on age/sex (within 7 days prior to start of protocol therapy) Age: Maximum serum creatinine (mg/dL)

  1 month to < 6 months: 0.4 mg/dL (male); 0.4 mg/dL (female) 6 months to < 1 year: 0.5 mg/dL (male); 0.5 mg/dL (female)

  1 to < 2 years: 0.6 mg/dL (male); 0.6 mg/dL (female) 2 to < 6 years: 0.8 mg/dL (male); 0.8 mg/dL (female) 6 to < 10 years 1 mg/dL (male); 1 mg/dL (female) 10 to <13 years: 1.2 mg/dL (male); 1.2 mg/dL (female) 13 to < 16 years: 1.5 mg/dL (male); 1.4 mg/dL (female)

  ≥ 16 years: 1.7 mg/dL (male); 1.4 mg/dL (female)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age, and (within 7 days prior to start of protocol therapy)
* Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) ≤ 135 U/L* (within 7 days prior to start of protocol therapy)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Shortening fraction of ≥ 27% by echocardiogram, or
* Ejection fraction of ≥ 50% by radionuclide angiogram
* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months and T-cell count above the lower limit of normal are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

Exclusion Criteria:

* Patients who received prior radiotherapy to the head or neck
* Patients who received prior chemotherapy or radiation for the treatment of any cancer in the last 3 years. These patients must also be in remission
* Patients with a diagnosis of immunodeficiency
* Patients with an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive agents). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

  * Note: Patients with well-controlled asthma and no need for systemic steroids for the treatment of asthma in the last 12 months will not be excluded
* Patients with a condition requiring systemic treatment with either corticosteroids (> 0.25 mg/kg (10 mg) daily prednisone equivalent) within 14 days or other immunosuppressive medications within 30 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses > 0.25 mg/kg (10 mg) daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Patients with a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients with detectable viral load of human immunodeficiency virus (HIV), hepatitis B or hepatitis C, or active tuberculosis
* Patients who have undergone solid organ or allogeneic hematopoietic transplant at any time
* Due to risks of fetal and teratogenic adverse events as seen in animal studies, a negative pregnancy test must be obtained in females of childbearing potential, defined as females who are post-menarchal. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Females of childbearing potential that are sexually active must agree to either practice 2 medically accepted highly-effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 5 months after the last dose of nivolumab, 6 months after the last dose of gemcitabine, and 14 months after the last dose of cisplatin, whichever is longer
* Males of childbearing potential that are sexually active must agree to either practice a medically accepted highly-effective methods of contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 3 months after the last dose of gemcitabine, and 11 months after the last dose of cisplatin, whichever is longer
* Lactating females are not eligible unless they have agreed not to breastfeed their infants starting with the first dose of study therapy through 5 months after the last dose of nivolumab
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher immune-related adverse events (irAE) during induction chemoimmunotherapy (CIT) | Until the end of consolidation therapy
  Will be assessed by Common Terminology Criteria for Adverse Events. IrAEs include diarrhea (noninfectious), colitis (noninfectious), pneumonitis (noninfectious), myocarditis, elevated alanine aminotransferase, elevated aspartate aminotransferase, pancreatitis, elevated blood bilirubin, hypophysitis and hyperthyroid considered possibly, probably, or definitely related to nivolumab.

SECONDARY OUTCOMES:
Event-free survival (EFS) | From date of enrollment to the earliest occurrence of date of relapse, disease progression, second malignant neoplasm or death due to any cause, assessed at 2 years
  EFS along with the 95% confidence intervals will be estimated using the Kaplan-Meier method. The EFS will be reported separately for patients with non-metastatic disease and those with metastatic disease (if there are enough patients with metastatic disease enrolled).
Objective response rate | At the end of induction CIT
  Will be defined as the rate of responders among evaluable patients using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Feasibility success of the induction regimen | At the end of induction CIT
  Will be defined as the completion of three cycles of induction without delay of greater than 30 days for radiation initiation due to toxicity in 80% of patients.
Cumulative incidence of local or distant relapse | Up to 5 years
  Defined as a function of time since enrollment will be estimated by the method of Gray.

OTHER OUTCOMES:
EFS | At 5 years
  Will be assessed using Kaplan-Meier estimates.
Overall survival | From date of enrollment to death due to any cause or date of last follow-up, assessed at 5 years
  Will be assessed using Kaplan-Meier estimates.
Proportion of patients who achieve complete response | At the end of induction and maintenance
  Will be assessed by retrospective central review by the proportion of patients who achieve complete response by magnetic resonance imaging using RECIST 1.1 criteria and the proportion of patients who achieve complete metabolic response using Positron Emission Tomography Response Criteria In Solid Tumors criteria at the end of induction and the end of maintenance based on central review will be presented. A two-way table of response assessments according to the two modalities will be constructed and McNemar's test will be performed to evaluate the concordance.
Protocol deviation related to radiation therapy delivery | Up to 5 years
  Will be assessed by retrospective central review. The effect of deviation, categorized as present or absent by the central reviewer, on the hazard of EFS will be estimated by Cox proportional hazard model. The hazard ratio will be reported along with 95% confidence interval.
EFS in patients receiving intensity modulated radiation therapy with those who receive proton therapy | Up to 5 years
  Will be assessed using a log-rank test.
Incidence of grade 3 or higher adverse events | Up to 5 years
  Will be assessed during protocol therapy. The incidence of these events will be reported for each toxicity term. Furthermore, the irAE and toxicity related to radiation will be summarized by toxicity term and will be presented separately for the on-protocol therapy period and long-term follow-up.
Swallowing dysfunction | At baseline, during induction prior to start of chemoradioimmunotherapy (CRIT), each cycle throughout CRIT, within 3 months after maintenance and yearly at follow up, up to 5 years
  Will be assessed using modified Functional Oral Intake Scale (FOIS) and pediatric Eating Assessment Tool (EAT)-10. The EAT-10 consists of 10 items scored from 0 (no impairment) to 4 (severe impairment). Total scores range from 0 to 40; higher scores indicate greater self-perceived impairment. Modified FOIS is an ordinal scale is a rating scale with 7 points for adults and 5 points in pediatrics. It is used to describe the feeding status and patients with dysphagia. Level 1 indicates inability to take anything by mouth while the highest point indicates full oral feeding. Will summarize responses from the modified FOIS and pediatric EAT-10 descriptively for each of these time points. A two-sided Wilcoxon rank-sum test will be performed to test the null hypothesis of equal score between two groups (who receive 54Gy versus 59.4Gy) at the end of the CRIT. Will evaluate the potential impact of other factors, as appropriate, such as baseline scores or disease stages for this analysis.
Quality of life | At baseline, during induction prior to start of CRIT, each cycle throughout CRIT, within 3 months after maintenance and yearly at follow up, up to 5 years
  Will be assessed using Patient-Reported Outcomes Measurement Information System (PROMIS). PROMIS includes multiple measures such as physical function mobility, anxiety, depressive symptoms, fatigue, etc. PROMIS use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation of that population. Higher T-score indicates more of the concept being measured. The numerical T scores of each domain will be summarized descriptively at every time point.
Lymphocyte-to-monocyte ratio (LMR) | At baseline, pre-radiation/consolidation, and post-radiation pre-maintenance
  Will be assessed the ratio calculated by dividing the absolute lymphocyte count by the absolute monocyte count from a complete blood count with differential analysis performed. Lymphocyte and monocyte counts will be collected at the following time points: baseline, pre-radiation/consolidation, and post-radiation pre-maintenance. Cox proportional hazards regression will be used to evaluate the association between baseline LMR and EFS. The hazard ratio will be reported with a 95% confidence interval. In addition, the LMR will be summarized descriptively by the evaluation time points.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn D Gartrell, Principal Investigator — Children's Oncology Group
Locations (81):
- United States (73):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- University Pediatric Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm